CLINICAL TRIAL: NCT04750954
Title: A Phase 1b Trial of M3814 (Peposertib) in Combination With Lutetium 177 Dotatate for Well-Differentiated Somatostatin Receptor-Positive Gastroenteropancreatic Neuroendocrine Tumors (GEP-NETs)
Brief Title: Testing the Addition of An Anti-cancer Drug, M3814 (Peposertib), to the Usual Radiation-Based Treatment (Lutetium Lu 177 Dotatate) for Pancreatic Neuroendocrine Tumors
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2021-00860; NCI-2021-00860 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10450-36MTC; 10450 (Other: Ohio State University Comprehensive Cancer Center LAO); 10450 (Other: CTEP); UM1CA186712 (NIH)
Record Dates: First submitted 2021-02-10; First posted 2021-02-11 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Neuroendocrine Neoplasm
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — Specimen Handling; lutetium Lu 177 dotatate; Magnetic Resonance Spectroscopy; peposertib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (peposertib, lutetium Lu 177 dotatate) (Experimental): Patients receive peposertib PO QD or BID on days 1-21 and lutetium Lu 177 dotatate IV over 30 minutes on day 1. Treatment repeats every 56 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo CT/MRI throughout the trial and undergo collection of blood samples on study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Drug: Lutetium Lu 177 Dotatate; Procedure: Magnetic Resonance Imaging; Drug: Peposertib

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Drug: Lutetium Lu 177 Dotatate — Given IV
  Other Names: 177 Lu-DOTA-TATE; 177 Lu-DOTA-Tyr3-Octreotate; 177Lu-DOTA0-Tyr3-Octreotate; Lutathera; Lutetium (177Lu) Oxodotreotide; Lutetium Lu 177 DOTA(0)-Tyr(3)-Octreotate; Lutetium Lu 177-DOTA-Tyr3-Octreotate; lutetium Lu 177-DOTATATE; Lutetium Oxodotreotide Lu-177
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Drug: Peposertib — Given PO
  Other Names: 3-Pyridazinemethanol, alpha-(2-Chloro-4-fluoro-5-(7-(4-morpholinyl)-4-quinazolinyl)phenyl)-6-methoxy-, (alphaS)-; M 3814; M-3814; M3814; MSC 2490484A; MSC-2490484A; MSC2490484A; Nedisertib

SUMMARY:
This phase Ib trial is to find out the best dose, possible benefits and/or side effects of peposertib when given together with lutetium Lu 177 dotatate in treating patients with neuroendocrine tumors. Peposertib may stop the growth of tumor cells by blocking some of the enzymes needed for cell formation, so as to help block the formation of growths that may become cancer. Radioactive drugs, such as lutetium Lu 177 dotatate, may deliver radiation directly to tumor cells and not harm normal cells. Adding peposertib to lutetium Lu 177 dotatate may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the safety and to determine the recommended phase 2 dose (RP2D) of lutetium Lu 177 dotatate in combination with M3814 (peposertib).

SECONDARY OBJECTIVES:

I. To observe and record anti-tumor activity. II. To determine the overall response rate (ORR) by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 at 4, 8, and 12 months post-therapy.

III. To measure duration of response (DOR) associated with the combination. IV. To evaluate progression-free survival (PFS).

CORRELATIVE OBJECTIVES:

I. Measure the somatostatin receptor uptake on gallium 68 dotatate or Copper 64 dotatate at baseline.

II. Perform lutetium Lu 177 dotatate dosimetry. III. Determine the pharmacokinetic (PK) parameters of M3814 (peposertib). IV. Describe the tumor molecular profile using whole exome sequencing (WES) and ribonucleic acid (RNA) sequencing (RNAseq) and correlate it with treatment outcome.

V. Collect plasma for circulating tumor deoxyribonucleic acid (DNA) (ctDNA) assessment.

VI. Collect blood for biobanking and future correlative studies. VII. Measure association of overall response rate with gallium 68 dotatate-positron emission tomography (PET)/computed tomography (CT) or Copper 64 dotatate measurements and Krenning score.

OUTLINE: This is a dose-escalation study of peposertib followed by a dose-expansion study.

Patients receive peposertib orally (PO) once daily (QD) or twice daily (BID) on days 1-21 and lutetium Lu 177 dotatate intravenously (IV) over 30 minutes on day 1. Treatment repeats every 56 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo CT/magnetic resonance imaging (MRI) throughout the trial and undergo collection of blood samples on study.

After completion of study treatment, patients are followed up every 4 months for 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed well-differentiated neuroendocrine tumor with positive dotatate scan (gallium 68 or copper 64) (as determined by the site principal investigator [PI]) within 6 months before enrollment. Lesions on the dotatate scan (gallium 68 or copper 64) are considered positive if the maximum standard uptake value (SUVmax) is > 2 times the mean standard uptake value (SUVmean) of normal liver parenchyma. Patients must have the gallium 68 or copper 64 dotatate scans available to send for central review before enrollment
* Patients must have measurable progressive disease based on RECIST criteria, version 1.1, evidenced with CT/MRI scans obtained within 12 months before enrollment
* Failure of at least one prior systemic cancer treatment with somatostatin analogs
* No prior exposure to peptide receptor radionuclide therapy
* Age >= 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* White blood cell count >= 2,000/mcL
* Absolute neutrophil count >= 1,000/mcL
* Platelets >= 75,000/mcL
* Hemoglobin >= 8.0 g/dL
* Total bilirubin =< 1.5 x institutional upper limit of normal (ULN)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) =< 3 x institutional ULN
* Alkaline phosphatase =< 3 x institutional ULN
* Glomerular filtration rate (GFR) >= 50 mL/min/1.73 m^2 (per the Cockcroft-Gault [C-G])
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class 2B or better
* Patients must have recovered from adverse events of previously administered therapeutic agents to grade 2 or less toxicity according to Common Terminology Criteria for Adverse Events (CTCAE) 5.0
* Pregnancy Precaution: Women should avoid pregnancy for seven months after the date of their last treatment with lutetium Lu 177 dotatate. Men should avoid fathering a child for 4 months after the last dose of Lutetium Lu 177 dotatate. It is noteworthy that beta-human chorionic gonadotropin (HCG) may be secreted by a small percentage of neuroendocrine tumor (NET)s, such that, in addition to being a pregnancy marker, it also is a tumor marker. Consequently, NET female patients with positive beta-HCG (> 5 mIU/mL) at baseline can be eligible to enter the study and receive treatment if pregnancy can be excluded by lack of expected doubling of beta-HCG and negative pelvic ultrasound. Normally, in pregnant subjects beta-HCG doubles every 2 days during the first 4 weeks of pregnancy and every 3.5 days by Weeks 6 to 7. Women of childbearing potential include any female who has experienced menarche and who has not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation, or bilateral ovariectomy) or is not postmenopausal (defined as amenorrhea > 12 consecutive months, and for women on hormone replacement therapy, only with a documented plasma follicle-stimulating hormone [FSH] level > 35 mIU/mL). Even women who are using oral, implanted, or injected contraceptive hormones, an intrauterine device (IUD), or barrier methods (diaphragm, condoms, spermicidal) to prevent pregnancy, are practicing abstinence, or where the partner is sterile (e.g., vasectomy) should be considered to be of childbearing potential. Postmenopausal women who have fertilized eggs implanted are also considered to be of childbearing potential. Acceptable methods of contraception may include total abstinence at the discretion of the Investigator in cases where the age, career, lifestyle, or sexual orientation of the patient ensures compliance. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception. Reliable contraception (hormonal or barrier method of birth control; abstinence) should be maintained throughout the study and for 7 months after study treatment discontinuation, for women, and for 4 months for men. All women of childbearing potential and male partners must use a double-barrier method of birth control or practice continuous abstinence from heterosexual contact throughout the study and for seven months after the end of the last treatment for women, and four months for men
* Ability to understand and the willingness to sign a written informed consent document. Participants with impaired decision-making capacity (IDMC) who have a legally-authorized representative (LAR) and/or family member available will also be eligible.

Exclusion Criteria:

* Patients who have had major surgical procedures in the 4 weeks prior to enrollment
* Patients are excluded if they received prior systemic peptide receptor radionuclide therapy (PRRT)-based therapies
* Patients with an inability to swallow oral medications or gastrointestinal disease limiting absorption of oral agents
* Patients who are receiving any other investigational agents
* Known brain metastases, unless these metastases have been treated and stabilized for at least 4 weeks, prior to enrollment in the study. Patients with a history of brain metastases must have either a head CT with contrast or brain MRI to document stable disease prior to enrollment in the study
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to M3814 (peposertib) or lutetium Lu 177 dotatate
* Prior external beam radiotherapy to more than 50% of bone marrow (whole body) will be excluded, as determined by a radiation medicine physicist who will calculate the volume of bone marrow exposure in prior radiotherapy portals divided by the volume of total bone marrow harboring tissues. This ratio must be less than 50 percent
* Patients who cannot discontinue concomitant medications or herbal supplements that are strong inhibitors or strong inducers of cytochrome P450 (CYP) isoenzymes CYP3A4/5, CYP2C9, and CYP2C19. Concomitant use of CYP3A4/5, 1A2, 2B6, 2C8, substrates with a narrow therapeutic index are also excluded. Patients may confer with the study doctor to determine if alternative medications can be used. The following categories of medications and herbal supplements must be discontinued for at least the specified period of time before the patient can be treated:

  * Strong inducers of CYP3A4/5, CYP2C9 and CYP2C19: >= 3 weeks prior to study treatment
  * Strong inhibitors of CYP3A4/5, CYP2C9 and CYP2C19: >= 1 week prior to study treatment
  * Substrates of CYP3A4/5, 1A2, 2B6, 2C8, with a narrow therapeutic index: >= 1 day prior to study treatment Because the lists of these agents are constantly changing, it is important to regularly consult a frequently-updated medical reference. As part of the enrollment/informed consent procedures, the patient will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the patient is considering a new over-the-counter medicine or herbal product
* Patients who cannot discontinue concomitant proton-pump inhibitors (PPIs). Patients may confer with the study doctor to determine if such medications can be discontinued. These must be discontinued >= 5 days prior to study treatment. Patients do not need to discontinue calcium carbonate
* Patients with ongoing active infection or treatment with a live attenuated vaccine within 4 weeks of dosing. In addition, a negative polymerase chain reaction (PCR) test for Covid-19 infection is highly recommended before entering the study, and a close symptom follow up within the study
* Patients with uncontrolled intercurrent illness
* Patients with psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study because M3814 (peposertib) is a DNA-PK inhibitor and lutetium Lu 177 dotatate is a peptide receptor radionuclide therapy with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with M3814 (peposertib) and lutetium Lu 177 dotatate, breastfeeding should be discontinued if the mother is treated with M3814 (peposertib) and lutetium Lu 177 dotatate and for 2.5 months following the last lutetium Lu 177 dotatate treatment
* Discontinue long-acting somatostatin analogs (e.g., long-acting octreotide) for at least 4 weeks prior to initiating lutetium Lu 177 dotatate. Long-acting somatostatin analogs will be allowed to continue if patient has a history of carcinoid syndrome and requires long-acting somatostatin analogs for control of his/her functional syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2021-07-22 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Recommended phase 2 dose | Up to 8 weeks
Dose limiting toxicity | Up to 24 months post-treatment
  Will be assessed by Common Terminology Criteria for Adverse Events version 5.0. The maximum grade of toxicity for each adverse event category of interest will be recorded for each patient and the summary results will be tabulated by category and grade. Will describe all serious (>= grade 3) toxicity events on a patient-by-patient basis. Frequency and incidence tables of toxicity and adverse events will be generated in the overall patient group and by dose level depending on patient enrollment.

SECONDARY OUTCOMES:
Overall response rate | Up to 24 months post-treatment
  Will be estimated along with 95% exact binomial confidence interval.
Progression free survival | Up to 24 months post-treatment
  Will be estimated using the Kaplan-Meier curve and median estimates and confidence intervals will be calculated.
Overall survival | Up to 24 months post-treatment
  Will be estimated using the Kaplan-Meier curve and median estimates and confidence intervals will be calculated.

OTHER OUTCOMES:
Radiographic expression of somatostatin receptors | Baseline up to 24 months post-treatment
  Will be summarized using descriptive statistics and changes from baseline versus follow-up time points will be assessed using paired test methodologies.
Pharmacokinetic (PK) analysis | Baseline, cycle 1 days 2, 4, 9, 15, and 22
  PK parameters will be estimated from patients enrolled in the dose escalation portion of the phase 1 trial. PK parameters will be compared with historical controls, and exploratorily, may correlate exposure to toxicity, and incorporate data into a population PK model.
Krenning score from the gallium 68 or copper 64 dotatate | Up to 24 months post-treatment
  Will be summarized by calculating the proportion of patients in each Krenning score category and exploratory assessments for association with clinical response will be performed using Fisher's exact test. Median, interquartile range will be calculated for quantitative image measurements from gallium 68 or copper 64 dotatate and exploratory comparison of levels with clinical response will be performed using two sample t-test or nonparametric analogs.

CONTACTS AND LOCATIONS:
Overall Officials: Lowell B Anthony, Principal Investigator — Ohio State University Comprehensive Cancer Center LAO
Locations (5):
- United States (5):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm

REFERENCES:
- [Derived] Chauhan A, Prieur A, Kolesar J, Arnold S, Payen L, Mahi Y, Vire B, Sands M, Evers BM, Joubert D, Anthony L. hPG80 (Circulating Progastrin), a Novel Blood-Based Biomarker for Detection of Poorly Differentiated Neuroendocrine Carcinoma and Well Differentiated Neuroendocrine Tumors. Cancers (Basel). 2022 Feb 9;14(4):863. doi: 10.3390/cancers14040863. PMID 35205614

DOCUMENTS (1):
  • Informed Consent Form (2024-07-01): https://cdn.clinicaltrials.gov/large-docs/54/NCT04750954/ICF_000.pdf